CLINICAL TRIAL: NCT00834171
Title: A Retrospective Evaluation of the Intraocular Pressure Spikes With Loteprednol and Loteprednol/Tobramycin
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Vice President Medical Affairs, Allergan, Inc.
Other Study IDs: MA-RES-08-003
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-08

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Loteprednol Etabonate; Tobramycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 1: Loteprednol etabonate ophthalmic suspension 0.5%
  Interventions: Drug: Loteprednol etabonate ophthalmic suspension 0.5%
- 2: Loteprednol etabonate (0.5%) and tobramycin (0.3%)
  Interventions: Drug: Loteprednol etabonate (0.5%) and tobramycin (0.3%).

INTERVENTIONS:
Drug: Loteprednol etabonate ophthalmic suspension 0.5% — Apply one to two drops of Loteprednol etabonate ophthalmic suspension 0.5% into the conjunctival sac as prescribed by your physician
  Other Names: LOTEMAX®
  Groups: 1
Drug: Loteprednol etabonate (0.5%) and tobramycin (0.3%). — Apply one or two drops of Loteprednol etabonate (0.5%) and tobramycin (0.3%) into the conjunctival sac as prescribed by your physician.
  Other Names: Zylet®
  Groups: 2

SUMMARY:
Patient charts will be reviewed to evaluate the incidence of intraocular pressure spikes while on Loteprednol etabonate ophthalmic suspension 0.5%, Loteprednol etabonate (0.5%) and tobramycin (0.3%)

ELIGIBILITY:
Inclusion Criteria:

* Any patient who experienced an IOP spike while using Lotemax or Zylet will be included

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data to be collected will include: Patient Demographics (age, gender, race, eye color), medical and ophthalmic history, active ophthalmic disease, active systemic diseases, concomitant medications, procedure/condition for which Lotemax®/Zylet® were prescribed, underlying etiology requiring PK (if applicable), history of prior ocular surgery, prior history of steroid response, history of glaucoma, start/stop date of steroid treatment, IOP before and after steroid treatment, treatment-related adverse events, and any other notes/information that the investigator feels may be important.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Maclean, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Loteprednol Etabonate Ophthalmic Suspension 0.5%: Loteprednol etabonate ophthalmic suspension 0.5%
- Loteprednol Etabonate (0.5%) and Tobramycin (0.3%): Loteprednol etabonate (0.5%) and tobramycin (0.3%)
Period: Overall Study
Arm/Group | Loteprednol Etabonate Ophthalmic Suspension 0.5% | Loteprednol Etabonate (0.5%) and Tobramycin (0.3%)
Started | 43 | 7
Completed | 43 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate Ophthalmic Suspension 0.5% | Loteprednol Etabonate (0.5%) and Tobramycin (0.3%) | Total
Number analyzed (Participants) | 43 | 7 | 50
Age Continuous [Mean (Full Range); unit: years] | NA [NA to NA] — Baseline characteristics for age only analyzed for total study not for individual arms. | NA [NA to NA] — Baseline characteristics for age only analyzed for total study not for individual arms. | 58.8 [17 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — There were 33 females enrolled in the entire study. Baseline characteristics for gender only analyzed for total study not for individual arms. | NA — There were 33 females enrolled in the entire study. Baseline characteristics for gender only analyzed for total study not for individual arms. |
  Male | NA — There were 17 males enrolled in the entire study. Baseline characteristics for gender only analyzed for total study not for individual arms. | NA — There were 17 males enrolled in the entire study. Baseline characteristics for gender only analyzed for total study not for individual arms. |

OUTCOME MEASURES:

1. Primary Outcome: Mean Elevated Intraocular Pressure (IOP) During Treatment
Description: Mean elevated IOP during treatment. IOP is a measurement of the fluid pressure inside the eye. IOP was recorded any time an elevation of IOP (increase of 5 mmHg or more) occurred while using study treatment. The median duration of treatment at the time of observed IOP elevation was 55 days.
Time Frame: 55 days
Population: Intent to treat, which included all patients in the study.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Loteprednol Etabonate Ophthalmic Suspension 0.5% | Loteprednol Etabonate (0.5%) and Tobramycin (0.3%)
Number analyzed (Participants) | 43 | 7
Millimeters of mercury (mmHg) | 24.8 (6.9) | 23.9 (3.5)

ADVERSE EVENTS:
Arm/Group | Loteprednol Etabonate Ophthalmic Suspension 0.5% | Loteprednol Etabonate (0.5%) and Tobramycin (0.3%)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/7
Other Adverse Events (participants affected / at risk) | 4/43 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Loteprednol Etabonate Ophthalmic Suspension 0.5% (N=43) | Loteprednol Etabonate (0.5%) and Tobramycin (0.3%) (N=7)
Glaucoma surgery (Surgical and medical procedures) | 4 | 0 — Type of Glaucoma Surgery: * Baerveldt tube shunt (2 patients) * Cytophotocoagulation diode laser (1 patient) * Selective laser trabeculoplasty (1 patient)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo